CLINICAL TRIAL: NCT04967586
Title: Medical Students and Risk of COVID-19 Infection: a Descriptive Study From the University of Jordan
Brief Title: Medical Students and Risk of COVID-19 Infection
Acronym: Covid 19
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Amjad Bani Hani, Associate professor, University of Jordan
Other Study IDs: 2021/47
Record Dates: First submitted 2021-07-16; First posted 2021-07-19 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preclinical medical students
  Interventions: Other: No intervention, questioner only
- Clinical medical students
  Interventions: Other: No intervention, questioner only

INTERVENTIONS:
Other: No intervention, questioner only — questioner only

SUMMARY:
This study aims to estimate the prevalence of infected medical students with COVID-19 in the University of Jordan and to compare number of cases between students in clinical and basic years. In addition, this can provide insight into the awareness of infection control practices among students. Furthermore, to examine if hospital rotations increased risk of infection between clinical year medical students.

ELIGIBILITY:
Inclusion Criteria:

All medical Students

-

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical Students at The university of Jordan from second till sixth year
Sampling Method: Non-Probability Sample
Enrollment: 1830 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
COVID 19 infection | 3 months
  Incidence of Infected students with Covid 19

CONTACTS AND LOCATIONS:
Overall Officials: Amjad bani Hani, MD, Principal Investigator — The University of Jordan
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No